CLINICAL TRIAL: NCT03283774
Title: Multifactorial Control of Type 2 Diabetes and Treatment Intensity in Primary Care: A Cohort Study
Brief Title: Multifactorial Control of Type 2 Diabetes and Treatment Intensity in Primary Care
Acronym: eControl
Status: Completed | Type: Observational
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Other Study IDs: GOL-DML-2015-01
Record Dates: First submitted 2015-05-05; First posted 2017-09-14 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: current clinical practice — quality management (data registration, drug prescription, diagnostic and clinical tests ...), in primary care of patients with diabetes mellitus

SUMMARY:
Main Objective: To identify changes in metabolic control of type 2 diabetes in patients of the Catalan national health system during 2007-2013.

Study design: Follow-up of a population with type 2 diabetes during 7 years (2007-2013).

Study participants: Approximately 300,000 people with a clinical record in the SIDIAP database.

Source: SIDIAP database. Variables and measurements: Age, gender, time since diagnosis of type 2 diabetes, associated cardiovascular risk factors, micro- and macrovascular complications of diabetes, causes of mortality, treatment for hyperglycaemia and for modifiable risk factors, other conditions related to diabetes and its management. The economic costs of diabetes during the study period will also be analyzed.

Analysis: The clinical variables will be described and 95% confidence intervals will be calculated for the main variables associated with the study outcomes. Missing values will count as non-existing data and missing value imputation will not be used in the analysis. If a subgroup of patients is considered of particular interest, sub analyses will be carried out. Predictive variables of good metabolic control and of complications and mortality of diabetes will be analyzed with the hazard ratios for each factor.

Results:

Applicability: The results related to control of diabetes will serve as a basis for improving metabolic control and decreasing chronic complications and to optimize cost-effectiveness of treatments.

Significance: A long-term study of a population receiving usual treatment is required to understand the changes in indicators of metabolic control, morbidity and mortality and in the management of the disease.

Limitations: Those associated with the use of large population databases.

DETAILED DESCRIPTION:
Main Objective

• To determine the changes in metabolic control of type 2 diabetes during 2007-2013 in patients of the main Catalan public health provider (Catalan Health Service-CHS).

Secondary Objectives

* To describe changes in HbA1c values in the Catalan population with type 2 diabetes during 2007-2013.
* To describe changes and control of modifiable cardiovascular risk factors (blood pressure, lipid profile, smoking and obesity) in the Catalan population with type 2 diabetes during 2007-2013.
* To identify factors associated with changes in HbA1c and in the variables of metabolic control during the study period.
* To describe changes in the prevalence of macrovascular (ischemic heart disease, cerebrovascular accident, peripheral arterial disease) and microvascular complications (kidney disease, retinopathy) in the Catalan population with type 2 diabetes during 2007-2013.
* To describe changes in mortality in the Catalan population with type 2 diabetes during 2007-2013.
* To analyse the main costs of diabetes in Catalonia during 2007-2013.
* To describe changes in the use of hypoglycaemic agents in the Catalan population with type 2 diabetes during 2007-2013.
* To describe changes in the use of medicines to control cardiovascular risk factors (antihypertensive, hypolipidemic and antiplatelet agents) during 2007-2013.

Hypothesis During 2007-2013 the metabolic control of type 2 diabetes patients in the public health system of Catalonia (CHS) improves. The management of type 2 diabetes incorporates new pharmacological treatments.

Methods

Study Design Longitudinal study with cross-sectional, yearly analysis for each year of the study period (2007-2013).

Reference Population and Study Population A longitudinal study with a cross-sectional yearly analysis on June 30 of each year (DTALL) in those patients with a verified type 2 diabetes diagnosis will be carried out with SIDIAP data.

The observation period will be the calendar years 2007 (baseline), 2008, 2009, 2010, 2011, 2012 and 2013 (final).

The SIDIAP database includes the following information of the 5.8 million people from the 282 primary care centres of the Catalan Health Service linked with a unique, anonymized personal identifier:

1. Information from the electronic clinical records (eCAP): demographic data, visits to the primary care centre, health conditions (codes ICD-10), clinical variables, prescriptions, immunizations and referrals.
2. Blood tests results: will be directly retrieved from the laboratories databases.
3. Information on the medication dispensed in pharmacies: obtained from the pharmacy billing database of the Catalan Health Institute (CatSalut).

Data Collection and Information Sources The data sources are constituted by the electronic clinical records, blood tests results, the pharmacy register of the SIDIAP database and mortality data from AQuAS (Health Quality and Evaluation Agency of Catalonia)

Since the study does not target any specific treatment and no specific medication is considered an exposure therapy under investigation, no definition of exposure to any medication is included.

Data Analysis

Data analysis will be performed on study patients meeting inclusion criteria. The clinical variables will be described in terms of absolute and relative frequency for qualitative variables. Central tendency and dispersion measures will be used to describe quantitative variables as appropriate and 95% confidence intervals will be calculated for the main variables associated with the study outcomes.

Statistical tests will be used to compare the distribution of risk factors over time (DTALL): ANOVA will be used for normally distributed quantitative variables, the non-parametric equivalent (Kruskal-Wallis) will be used for non-normally distributed variables, and chi-square test will be used for categorical variables. The P value of the linear trend over the different time periods will be calculated for each variable. The cost associated with diabetes will be calculated for each time cohort.

The likelihood-ratio test will be used to test for interaction between the study variables (eg, HbA1c or cardiovascular events) in nested models with the terms of interaction included or removed. To analyse changes over time of variables to control diabetes in the study cohorts from 2007 to 2013, repeated measures ANCOVA and multinomial logistic regression analysis will be used for quantitative and categorical variables, respectively. These models will be then be adjusted for potential confounders.

The incidence rate per year will used to analyse the frequency of events during the follow-up period (eg. ischaemic heart disease, stroke). The Cox proportional hazard model will be adjusted for potential confounders. Linearity and risk proportionality will be graphically verified in every model using mean weighted residuals.

Missing values will count as non-existing data and missing value imputation will not be used in the analysis.

Statistical comparisons will be performed using two-tail hypothesis testing with level of significance of 0.05. Data management will be conducted by IDIAP Jordi Gol personnel using the SIDIAP database and data analysis will be conducted by epidemiologists and statisticians.

Study Limitations The main limitations of the study derive from the quality of the register of big databases. Previous studies with the SIDIAP showed the validity of most of the variables used in the current protocol.

Ethics

Confidentiality The study will follow the International Guidelines for Ethical Review of Epidemiological Studies (Council for the International Organizations of Medical Sciences -CIOMS-, Geneva, 1991), and the Declaration of Helsinki (revision 64th WMA General Assembly, Fortaleza, Brazil, October 2013).

The management, communication and transfer of data of the participants will comply with the Protection of Personal Data Organic Law of December 13, 15/1999.

Amendments in the study protocol will be communicated in writing to all investigators and to the appointed Clinical Research Ethics Committee (CREC) and to the competent authorities according to the order sas / 3470/2009.

Risk-benefit assessment The current study involves solely access to a database where the data are anonymized and unlinked. It does not carry therefore any risk for the patients.

Data Confidentiality All information in the SIDIAP database is anonymized and unlinked.

Use of electronic data Data extraction will be carried out from the SIDIAP electronic database.

Follow-up and final reports A final report with the results obtained will be reviewed and approved by the IDIAP Jordi Gol researchers. No interim reports are anticipated.

The report should be written following dates in the workplan; a copy of the report will be sent to the Clinical Research Ethics Committee that has authorised the study.

Conditions of Publication The results of this retrospective, observational study will be published in international journals with mention of the Clinical Research Ethics Committee and the sources of funding. None of the investigators will communicate to any third party the results of the study before final results and interpretation have been agreed.

Clinical Research Ethics Committee (CREC) The IDIAP Jordi Gol CREC will evaluate this study.

Conflict of Interests AstraZENECA will provide funding through a contract with the IDIAP Jordi Gol Foundation.

AstraZENECA will not interfere in data extraction, analysis and presentation of reports. The funding is unlinked to the results of the study.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients > 30 years of age with a clinical record in the SIDIAP database.
* Patients with a diagnosis of type 2 diabetes (codes ICD10: E11, E11.0-E11.9, E14, E14.0-E14.9) on June 30 (DTALL) of each year.

Exclusion Criteria:

* Patients with a diagnosis of type 1 diabetes (E10), gestational diabetes (O24), secondary diabetes (E12) or any other type of diabetes (E13)

Min Age: 31 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population is selected from 5,8 million people from the 282 primary care centres of the Catalan Health Service identified with an anonymized personal identifier and included in a unique patient registry called "SIDIAP" for primary care in Catalonia (North East region in Spain)
Sampling Method: Non-Probability Sample
Enrollment: 300000 (Actual)
Dates: Start 2015-01; Primary Completion 2015-04 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Diagnosis of the most common cardiovascular risk factors | 2007-2013
  High Blood Pressure (more then >140/90mm Hg), Dyslipidaemia, Smoking and Obesity
Level of of glycated haemoglobin (HbA1c) | 2007-2013
  The value closer and prior to the DTALL date will be considered. A window of up to a year before the DTALL date will be accepted (i.e., from July 1 of the previous year up to DTALL)
Average of the three last measurements of systolic and diastolic blood pressure | 2007-2013
  A window of up to a year before the DTALL date will be accepted (i.e., from July 1 of the previous year up to DTALL). If there are no 3 BP measurements, the average of 2 measurements or the value closer and prior to DTALL will be accepted
Levels of Total Cholesterol (TC), LDL Cholesterol (LDL-C), HDL Cholesterol (HDL-C), triglycerides (TGC) and non-HDL Cholesterol. | 2007-2013
  A window of up to a year before the DTALL date will be accepted (i.e., from July 1 of the previous year up to DTALL)
Body Mass Index (BMI) | 2007-2013
  A window of up to a year before the DTALL date will be accepted (i.e., from July 1 of the previous year up to DTALL). BMI values and calculation of BMI with weight in kg and height in m will be accepted. The height value accepted will be that closer to DTALL measured after 18 years of age. Priority will be given to the calculation with weight in kg and height in m over a BMI value. The date of the calculation of the BMI with the weight and height will determine the weight value
Kidney function: glomerular filtration estimated by MDRD | 2007-2013
  The value closer and prior to the DTALL date will be considered. A window of up to a year before the DTALL date will be accepted (i.e., from July 1 of the previous year up to DTALL)
Kidney function: urinary albumin excretion (albumin/creatinine ratio). | 2007-2013
  The value closer and prior to the DTALL date will be considered. A window of up to a year before the DTALL date will be accepted (i.e., from July 1 of the previous year up to DTALL)
Use of hypoglycaemic agents (oral and/or GLP1) and insulin on the DTALL date | 2007-2013
  Monotherapy and combined therapy with other hypoglycaemic agents will be analysed. Dosage will not be specified. Data of use will be obtained from the pharmacy billing of the Catalan Health Service (CatSalut).
Use of antihypertensive, hypolipidemic, antiplatelet and anticoagulant agents on the DTALL date | 2007-2013
  Monotherapy and therapy combined with hypoglycaemic agents will be analysed. Dosage will not be specified.
  Data of use will be obtained from the pharmacy billing of the Catalan Health Service (CatSalut)
Cardiovascular disease | 2007-2013
  Ischemic heart disese Cerebrovascular accident with codes Arterial peripheral disease with codes Heart failure with codes Cardiovascular procedures such as coronary revascularization, revascularization and non-traumatic lower extremity amputation
Diagnosis of Diabetic retinopathy | 2007-2013
  Diabetic retinopathy on the DTALL date
Causes of mortality in the population with type 2 diabetes during the study period | 2007-2013
  Causes of mortality in the population with type 2 diabetes during the study period
Cost analysis | 2007-2013
  Pharmacological treatment, which will include pharmacological treatment of diabetes complications.
  * Number of visits carried out by primary care professionals (physician, nurse and other)
  * Visits carried out by specialists.
  * Number of referrals.
  * Medical tests.
  * Sick leave days
  * Hospital admissions (number of days in hospital and cost)
  * Number of test strips used for self-monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Josep Franch, Principal Investigator — Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Locations (1):
- IDIAP Jordi Gol, Barcelona, Spain